CLINICAL TRIAL: NCT03476434
Title: Panchromoendoscopy for the Surveillance of Serrated Polyposis Syndrome, a Multicenter, Prospective and Randomized Trial.
Brief Title: Chromoendoscopy for Serrated Polyposis Syndrome
Acronym: SERRADA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universitario de Móstoles (Other)
Responsible Party: Principal Investigator, Jorge Lopez Vicente, Principal Investigator, Hospital Universitario de Móstoles
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: HUMostoles 29115
Record Dates: First submitted 2018-03-18; First posted 2018-03-26 (Actual); Last update posted 2018-03-27 (Actual); Status verified 2018-03

CONDITIONS: Colonic Polyp; Colonic Neoplasms; Colonic Cancer
Keywords: sessile serrated polyp; chromoendoscopy; indigo carmine
MeSH Terms: conditions — Colonic Polyps; Colonic Neoplasms

STUDY DESIGN:
Intervention Model Description: Patients are randomized into two groups with tandem explorations: in the group A or white light group (HR-WLE) where inspection is performed with white light in both colonoscopies, and in the group B or chromoendoscopy group (HR-CE) where a first inspection is performed with white light and the second with panchromoendoscopy with indigo carmine.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group A (HR-WLE) (No Intervention): Two tandem colonoscopies: first inspection was on high-resolution white-light endoscopy from the cecum/ileo-colonic anastomosis to the rectum, followed by a second inspection also on HR-WLE.
- group B (HR_CE) (Experimental): two tandem colonoscopies: first inspection was on HR-WLE from the cecum/ileo-colonic anastomosis to the rectum, followed by a second inspection with panchromoendoscopy on indigo carmine.
  Interventions: Device: chromoendoscopy with indigo carmine

INTERVENTIONS:
Device: chromoendoscopy with indigo carmine — the lumen of the colon is sprayed in a segmental fashion using 0.4% indigo carmine delivered via a specially designed dye spray catheter (Olympus PW-5V1) or via the accessory channel with a 50cc syringe filled with indigo carmine and air.
  Arms: group B (HR_CE)

SUMMARY:
Serrated polyposis syndrome (SPS) is the most common colorectal polyposis syndrome and is characterized by the combination of large and/or numerous serrated lesions (SLs) throughout the colorectum. SLs are classified into sessile serrated polyps (SSP) with or without dysplasia, hyperplastic polyps (HP) and traditional serrated adenomas (TSA). In 2010 the World Health Organization (WHO) defined this syndrome by any one of the following conditions: criterion I, at least 5 SLs proximal to the sigmoid colon with 2 or more of these being >10mm in size; criterion II, any SLs proximal to the sigmoid colon in a first-degree relative with SPS; criterion III, more than 20 SLs of any size distributed throughout the colon. It has been demonstrated that 11.8-28.5% of patients with SPS present with colorectal cancer (CRC) at diagnosis. Tandem colonoscopy studies have demonstrated that a significant number of lesions are missed during conventional colonoscopy. This finding is even more evident when focusing SLs where a 31% miss rate has been reported. SLs are often overlooked due to their typical appearance: flat morphology, similar colour to the surrounding mucosa, subtle and indistinctive borders. Chromoendoscopy (dye spraying onto the surface of the colon) enhances the detection of subtle and flat polyps in the colon. Until the date no studies have assessed the use of dye-based chromoendoscopy in SPS patients.

The aim of this trial was to evaluate the usefulness of panchromoendoscopy with indigo carmine for the detection of polyps in the colon in patients with SPS. Secondary aims were to estimate the SLs and adenoma miss rates in these patients.

Patients were randomized in a 1:1 distribution to one of the two arms of the study by a list of random numbers distributed by the coordinator center. After randomization, patients were submitted to tandem colonoscopies by the same endoscopist:

* In group A (HR-WLE) the first inspection was on high-resolution white-light endoscopy from the cecum/ileo-colonic anastomosis to the rectum, followed by a second inspection also on HR-WLE.
* In group B (HR-CE) the first inspection was on HR-WLE from the cecum/ileo-colonic anastomosis to the rectum, followed by a second inspection with panchromoendoscopy. For this, the lumen was sprayed in a segmental fashion using 0.4% indigo carmine delivered via a specially designed dye spray catheter (Olympus PW-5V1) or via the accessory channel with a 50cc syringe filled with indigo carmine and air. After allowing a few seconds for the dye to settle onto the mucosal surface, excess pools of indigo carmine were suctioned and the mucosa was then scrutinised.

Time to withdrawal from the cecum was measured using a stopwatch excluding time needed for polypectomy and biopsies.

Lesions detected during each inspection were described and then removed. Size (measured in comparison with an open biopsy forceps), morphology (using the Paris classification), location and polypectomy technique were recorded before removal. Histology was used as gold standard.

DETAILED DESCRIPTION:
Serrated polyposis syndrome (SPS) is the most common colorectal polyposis syndrome and is characterized by the combination of large and/or numerous serrated lesions (SLs) throughout the colorectum. SLs are classified into sessile serrated polyps (SSP) with or without dysplasia, hyperplastic polyps (HP) and traditional serrated adenomas (TSA). In 2010 the World Health Organization (WHO) defined this syndrome by any one of the following conditions: criterion I, at least 5 SLs proximal to the sigmoid colon with 2 or more of these being >10mm in size; criterion II, any SLs proximal to the sigmoid colon in a first-degree relative with SPS; criterion III, more than 20 SLs of any size distributed throughout the colon. It has been demonstrated that 11.8-28.5% of patients with SPS present with colorectal cancer (CRC) at diagnosis. Tandem colonoscopy studies have demonstrated that a significant number of lesions are missed during conventional colonoscopy. This finding is even more evident when focusing SLs where a 31% miss rate has been reported. SLs are often overlooked due to their typical appearance: flat morphology, similar colour to the surrounding mucosa, subtle and indistinctive borders. Chromoendoscopy (dye spraying onto the surface of the colon) enhances the detection of subtle and flat polyps in the colon. Until the date no studies have assessed the use of dye-based chromoendoscopy in SPS patients.

The aim of this trial was to evaluate the usefulness of panchromoendoscopy with indigo carmine for the detection of polyps in the colon in patients with SPS. Secondary aims were to estimate the SLs and adenoma miss rates in these patients.

Patients were randomized in a 1:1 distribution to one of the two arms of the study by a list of random numbers distributed by the coordinator center. After randomization, patients were submitted to tandem colonoscopies by the same endoscopist:

* In group A (HR-WLE) the first inspection was on high-resolution white-light endoscopy from the cecum/ileo-colonic anastomosis to the rectum, followed by a second inspection also on HR-WLE.
* In group B (HR-CE) the first inspection was on HR-WLE from the cecum/ileo-colonic anastomosis to the rectum, followed by a second inspection with panchromoendoscopy. For this, the lumen was sprayed in a segmental fashion using 0.4% indigo carmine delivered via a specially designed dye spray catheter (Olympus PW-5V1) or via the accessory channel with a 50cc syringe filled with indigo carmine and air. After allowing a few seconds for the dye to settle onto the mucosal surface, excess pools of indigo carmine were suctioned and the mucosa was then scrutinised.

Time to withdrawal from the cecum was measured using a stopwatch excluding time needed for polypectomy and biopsies.

Lesions detected during each inspection were described and then removed. Size (measured in comparison with an open biopsy forceps), morphology (using the Paris classification), location and polypectomy technique were recorded before removal. Histology was used as gold standard. Biopsies were processed and stained using standard methods, and were subsequently evaluated by experienced gastrointestinal pathologists in each center according to Vienna criteria of gastrointestinal epithelial neoplasia. Serrated lesions were classified according to the WHO 2010 classification into hyperplastic polyps, sessile serrated polyps, and traditional serrated adenomas. Cytological dysplasia among serrated polyps was analyzed both as presence/absence of dysplasia, as well as the presence of low-grade and high-grade dysplasia. Neoplastic extension vertically into the submucosal layer or beyond was classified as invasive cancer.All the procedures were done under superficial sedation (midazolam and/or fentanyl or pethidine) or under deep sedation with propofol at the discretion of the endoscopist. Procedures were performed with high definition systems [i.e: 180/190 series in combination with EVIS EXERA II-III processors (Olympus, Tokyo, Japan), EC 390 LI scope in combination with Pentax processor (Pentax, Tokyo, Japan) or 590 WL and 580 ZW endoscopes in combination with Fujinon 4400/4450 processors (Fujifilm medical systems, USA)].

Quality of bowel cleansing was graded by each endoscopist following the Boston Bowel Preparation Scale. Adequate preparation was defined as a total score ≥6 with no segments <2. Procedures in which the quality of preparation was inadequate were excluded.

Sample size calculation: a polyp miss rate of 29% with HR-WLE was described previously in a Dutch multicenter study with SPS patients. Estimating a power of 80% and a significance level of 0.05, the investigators calculated 516 lesions would be required to measure a difference of 15% on HR-CE. In a previous study a median of 6 polyps was found on annual surveillance4. The investigators calculated a simple size of 86 patients for the study, 43 on each group.

Statistical analysis was performed with SPSS version 15.0 for windows. Numeric variables are presented as mean and standard deviation in case of a normal distribution and compared with a Student´s t test. Categorical variables are presented as frequencies and compared with the Chi Square test. Polyp miss rates were compared with chi square test. Logistic regression analysis was used to compare polyp characteristics and miss rates and was expressed as Odds ratio with the confidence intervals (95% CIs) to quantify the magnitude of the associations.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Serrated Polyposis Syndrome aged 18 years or older, fulfilling WHO criteria I or III.
* Clearing of all polyps previously achieved. Polyp "clearing" considered when all polyps >3 mm were removed during previous colonoscopies and/or partial colonic surgery when needed.
* Surveillance colonoscopy.

Exclusion Criteria:

* Inflammatory bowel disease.
* Hereditary CRC syndromes (i.e, APC, MUTYH - biallelic - and MMR genes germline mutations).
* Total colectomy.
* Decline for participation.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2015-02 (Actual); Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
polyp miss rate | through study completion, an average of 2 years
  number of polyps detected during the second inspection divided by the total number of polyps detected during the first and the second examination

SECONDARY OUTCOMES:
serrated lesions miss rate | through study completion, an average of 2 year
  number of serrated lesions detected during the second inspection divided by the total number of serrated lesions detected during the first and the second examination
adenoma miss rate | through study completion, an average of 2 year
  number of adenomas detected during the second inspection divided by the total number of adenomas detected during the first and the second examination

CONTACTS AND LOCATIONS:
Overall Officials: Jorge Lopez Vicente, Principal Investigator — Hospital Universitario de Móstoles

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rubio CA, Stemme S, Jaramillo E, Lindblom A. Hyperplastic polyposis coli syndrome and colorectal carcinoma. Endoscopy. 2006 Mar;38(3):266-70. doi: 10.1055/s-2006-925026. PMID 16528654
- [Background] East JE, Saunders BP, Jass JR. Sporadic and syndromic hyperplastic polyps and serrated adenomas of the colon: classification, molecular genetics, natural history, and clinical management. Gastroenterol Clin North Am. 2008 Mar;37(1):25-46, v. doi: 10.1016/j.gtc.2007.12.014. PMID 18313538
- [Background] Gao Q, Tsoi KK, Hirai HW, Wong MC, Chan FK, Wu JC, Lau JY, Sung JJ, Ng SC. Serrated polyps and the risk of synchronous colorectal advanced neoplasia: a systematic review and meta-analysis. Am J Gastroenterol. 2015 Apr;110(4):501-9; quiz 510. doi: 10.1038/ajg.2015.49. Epub 2015 Mar 10. PMID 25756237
- [Result] Boparai KS, Mathus-Vliegen EM, Koornstra JJ, Nagengast FM, van Leerdam M, van Noesel CJ, Houben M, Cats A, van Hest LP, Fockens P, Dekker E. Increased colorectal cancer risk during follow-up in patients with hyperplastic polyposis syndrome: a multicentre cohort study. Gut. 2010 Aug;59(8):1094-100. doi: 10.1136/gut.2009.185884. Epub 2009 Aug 25. PMID 19710031
- [Result] Carballal S, Rodriguez-Alcalde D, Moreira L, Hernandez L, Rodriguez L, Rodriguez-Moranta F, Gonzalo V, Bujanda L, Bessa X, Poves C, Cubiella J, Castro I, Gonzalez M, Moya E, Oquinena S, Clofent J, Quintero E, Esteban P, Pinol V, Fernandez FJ, Jover R, Cid L, Lopez-Ceron M, Cuatrecasas M, Lopez-Vicente J, Leoz ML, Rivero-Sanchez L, Castells A, Pellise M, Balaguer F; Gastrointestinal Oncology Group of the Spanish Gastroenterological Association. Colorectal cancer risk factors in patients with serrated polyposis syndrome: a large multicentre study. Gut. 2016 Nov;65(11):1829-1837. doi: 10.1136/gutjnl-2015-309647. Epub 2015 Aug 11. PMID 26264224
- [Result] Hazewinkel Y, Lopez-Ceron M, East JE, Rastogi A, Pellise M, Nakajima T, van Eeden S, Tytgat KM, Fockens P, Dekker E. Endoscopic features of sessile serrated adenomas: validation by international experts using high-resolution white-light endoscopy and narrow-band imaging. Gastrointest Endosc. 2013 Jun;77(6):916-24. doi: 10.1016/j.gie.2012.12.018. Epub 2013 Feb 21. PMID 23433877
- [Result] Hazewinkel Y, Tytgat KM, van Leerdam ME, Koornstra JJ, Bastiaansen BA, van Eeden S, Fockens P, Dekker E. Narrow-band imaging for the detection of polyps in patients with serrated polyposis syndrome: a multicenter, randomized, back-to-back trial. Gastrointest Endosc. 2015 Mar;81(3):531-8. doi: 10.1016/j.gie.2014.06.043. Epub 2014 Aug 1. PMID 25088921
- [Result] Boparai KS, van den Broek FJ, van Eeden S, Fockens P, Dekker E. Increased polyp detection using narrow band imaging compared with high resolution endoscopy in patients with hyperplastic polyposis syndrome. Endoscopy. 2011 Aug;43(8):676-82. doi: 10.1055/s-0030-1256447. Epub 2011 Aug 2. PMID 21811939
- [Result] Kaminski MF, Hassan C, Bisschops R, Pohl J, Pellise M, Dekker E, Ignjatovic-Wilson A, Hoffman A, Longcroft-Wheaton G, Heresbach D, Dumonceau JM, East JE. Advanced imaging for detection and differentiation of colorectal neoplasia: European Society of Gastrointestinal Endoscopy (ESGE) Guideline. Endoscopy. 2014 May;46(5):435-49. doi: 10.1055/s-0034-1365348. Epub 2014 Mar 17. PMID 24639382
- [Derived] Lopez-Vicente J, Rodriguez-Alcalde D, Hernandez L, Riu Pons F, Vega P, Herrero Rivas JM, Santiago Garcia J, Salces Franco I, Bustamante Balen M, Lopez-Ceron M, Pellise M; Endoscopy for High Risk Cancer Conditions group of the Spanish Gastroenterological Association and Spanish Digestive Endoscopy Society. Panchromoendoscopy Increases Detection of Polyps in Patients With Serrated Polyposis Syndrome. Clin Gastroenterol Hepatol. 2019 Sep;17(10):2016-2023.e6. doi: 10.1016/j.cgh.2018.10.029. Epub 2018 Oct 24. PMID 30366156